CLINICAL TRIAL: NCT02810743
Title: Substantially Improving the Cure Rate of High-risk BRCA1-like Breast Cancer Patients With Personalized Therapy (SUBITO) - an International Randomized Phase III Trial
Brief Title: Substantially Improving the Cure Rate of High-risk BRCA1-like Breast Cancer
Acronym: Subito
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16BRC
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Stage III; HER2 negative; homologous recombination deficiency (HRD)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ddAC-CP-Olaparib (Active Comparator): ddAC; doxorubicin 60 mg/m² as an i.v. bolus and cyclophosphamide 600 mg/m² as an i.v. bolus on day 1 every 2 weeks ddAC must be supported with prophylactic pegfilgrastim 6 mg s.c. given 24-48 hours after completion of administration of EVERY chemotherapy cycle
  CP; carboplatin/paclitaxel (CP) consisting of carboplatin (AUC 6) on day 1 and paclitaxel (80 mg/m2) on day 1,8 and 15 of a 21 days cycle. In total 4 courses of CP will be administered.
  Olaparib will be administered in Dutch centers only, as monotherapy for one year at a dose of 300 mg BID, starting 3 weeks after adjuvant radiotherapy, or, if radiotherapy is not indicated, 3-5 weeks after the last CP cycle.
  Patients without a (near) pCR will receive adjuvant capecitabine at a starting dose of 1000-1250 mg/m2, twice a day, on days 1-14 every 3 weeks for eight cycles.
  Interventions: Drug: ddAC-CP-Olaparib
- ddAC-mini CTC (Active Comparator): ddAC; doxorubicin 60 mg/m² as an i.v. bolus and cyclophosphamide 600 mg/m² as an i.v. bolus on day 1 every 2 weeks ddAC must be supported with prophylactic pegfilgrastim 6 mg s.c. given 24-48 hours after completion of administration of EVERY chemotherapy cycle
  intensified alkylating 'mini' CTC (2x) cyclophosphamide 3000 mg/m2 day 1 mesna 500 mg (push) + 2000 mg in 24 hours day 1 carboplatin (400 mg/m2; (or AUC=5 in patients with a calculated creatinine-clearance of <100 ml/min)) days 1,2 thiotepa 250 mg/m2 day 2
  Patients without a (near) pCR will receive adjuvant capecitabine at a starting dose of 1000-1250 mg/m2, twice a day, on days 1-14 every 3 weeks for eight cycles.
  Interventions: Drug: ddAC-mini CTC

INTERVENTIONS:
Drug: ddAC-CP-Olaparib — ddAC-CP-Olaparib
  Arms: ddAC-CP-Olaparib
Drug: ddAC-mini CTC — ddAC - mini CTC
  Arms: ddAC-mini CTC

SUMMARY:
Investigator-initiated, international, multicentre, randomized, open-label, (neo)adjuvant phase III study in target population (stage III, HER2-negative, BRCA1-like breast cancer patients) comparing optimized standard-dose chemotherapy with intensified, alkylating chemotherapy with stem cell rescue.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with stage III adenocarcinoma of the breast harboring signs of a breast cancer with features of homologous recombination deficiency (HRD)
* Age of 18-65 years
* The tumor must be HER2-negative
* Treatment must start within 8 weeks after the last surgical resection
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Previous radiation therapy
* Previous chemotherapy
* Any previous treatment with a PARP-inhibitor, including olaparib
* Pre-existing neuropathy from any cause in excess of Grade 1
* Chronic concomitant use of known strong or moderate CYP3A inducers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2033-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival in all patients | assessed up to 120 months
  time from randomization to death from any cause in all patients

SECONDARY OUTCOMES:
Overall survival in patients without a germline BRCA1/2 mutation | assessed up to 120 months
  time from randomization to death from any cause in without a germline BRCA1/2 mutation
Recurrence free interval in all patients | assessed up to 120 months
  time from randomization to local recurrence, second primary, distant recurrence or death, whichever comes first in all patients
Recurrence free interval in patients with an HR impaired tumor | assessed up to 120 months
  time from randomization to local recurrence, second primary, distant recurrence or death, whichever comes first in patients with an HR impaired tumor
Incidence of toxicity, graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.03 | up to 30 days after end of treatment
  Incidence of toxicity, graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.03
cost-effectiveness measured by costs per quality-adjusted life years (QALYs) | assessed up to 120 months
  cost-effectiveness measured by costs per quality-adjusted life years (QALYs)
Patient reported outcomes | assessed up to 24 months
  Patient reported outcomes; including quality of life (QoL) determined by a comprehensive panel of QoL questionnaires
cost-effectiveness measured by incremental cost-effectiveness ratio (ICER) | assessed up to 120 months
  cost-effectiveness measured by incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Linn, Prof. MD, Principal Investigator — NKI-AvL
Locations (11):
- France (2):
  - Institut Paoli Calmettes, Marseille
  - Hopital Tenon, University Marie-Curie, Paris
- Netherlands (9):
  - Medical spectrum Twente, Enschede, Overijssel
  - Antoni van Leeuwenhoek, Amsterdam
  - AZVU, Amsterdam
  - University Medical Center Groningen, Groningen
  - LUMC, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud UMC, Nijmegen
  - Erasmus Medical Center Cancer Institute, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided